CLINICAL TRIAL: NCT00994305
Title: Protective Effect of N-acetylcysteine on Early Outcomes of Deceased Renal Transplant
Acronym: NACTX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: ANTONIO MARMO LUCON, University of Sao Paulo Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NACTX; FAPESP 06/52046-0; CAPPesq 076/05
Record Dates: First submitted 2009-10-09; First posted 2009-10-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Renal Transplantation
Keywords: kidney transplantation; oxidative stress; acetylcysteine; graft rejection
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetylcysteine (Active Comparator): N-acetylcysteine 600 mg bid po 0-7 PO
  Interventions: Drug: N-acetylcysteine
- control (Sham Comparator): No treatment: standard care provided. No N-acetylcysteine administration.
  Interventions: Drug: control

INTERVENTIONS:
Drug: N-acetylcysteine — 600 mg bid po 0-7 PO
  Other Names: Fluimucil
  Arms: N-acetylcysteine
Drug: control — No treatment: standard care provided. No N-acetylcysteine administration.
  Other Names: N/A (not applicable)
  Arms: control

SUMMARY:
Investigate the therapeutic effects of the antioxidant N-acetylcysteine on early outcomes of deceased renal transplant patients.

DETAILED DESCRIPTION:
Investigate the therapeutic effects of 600 mg bid po of N-acetylcysteine on early outcomes of deceased renal transplant patients regarding oxidative stress and renal function.

Adult primary graft recipients of deceased renal donors will be randomly assign to treatment (NAC) or control group and prospectively evaluated for 90 days. Treatment group will receive N-acetylcysteine 600 mg bid po from 0 to 7th postoperative day (PO). Renal function will be determined by serum creatinine, Cockroft-Gault estimated GFR (eGFR) at 7th, 15th, 30th, 60th and 90th PO and dialysis free Kaplan-Meier estimate curve. Serum levels of thiobarbituric acid reactive substances (TBARS), which are markers of lipid peroxidation and oxidative stress, will be determined using the thiobarbituric acid assay from 0-7th PO. Statistical analysis will be performed using SPSS 16.0.

ELIGIBILITY:
Inclusion Criteria:

* primary deceased renal transplant recipients
* adult (>18 yo)

Exclusion Criteria:

* unable to drink N-acetylcysteine during the first 7 PO
* participation in other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2005-04; Primary Completion 2008-06 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress: measure of the oxidative stress generated after the deceased renal transplant by laboratorial serum measure of Thiobarbituric Acid Reactive Substances (TBARS) with the Trichloroacetic acid method. | 7 days

SECONDARY OUTCOMES:
Graft function: measure of serum creatinine | 3 months
Graft function:estimated creatinine clearance by Cokcroft-Gault formula | 3 months
Graft function: dialysis free status by Kaplan-Meier actuarial curve of recipients free from dialysis after deceased renal transplant | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Danilovic, MD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital Kidney Transplant Unit, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Danilovic A, Lucon AM, Seguro AC, Shimizu MHM, Ianhez LE, Nahas WC, Srougi M. N-acetylcysteine attenuates oxidative stress in deceased renal transplantation. The Journal of Urology 181 (4): 740; 2009.